CLINICAL TRIAL: NCT02166450
Title: Effects of Denture-Related Stomatitis on Blood Pressure, Endothelial Function and Systemic Immune Response in Patients With Dentures
Brief Title: Effects of Denture-Related Stomatitis on Blood Pressure in Denture Wearers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Guzik, MD, PhD, Jagiellonian University
Other Study IDs: DRS-001
Record Dates: First submitted 2014-06-13; First posted 2014-06-18 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Denture Stomatitis
Keywords: Denture stomatitis; Dentures; Denture wearers
MeSH Terms: conditions — Stomatitis, Denture | interventions — Nystatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Denture wearers without clinical signs of denture-related stomatitis confirmed with negative Candida swabs.
- Denture-related stomatitis group: Denture wearers with clinical signs of denture-related stomatitis, confirmed with positive Candida swabs.
  Treated for fungal infection, with nystatin [100 000 IU every 6 h for 3 weeks, applied on the infected area of the mucous membrane of the palate and cheeks].
  Interventions: Drug: Nystatin

INTERVENTIONS:
Drug: Nystatin — 100 000 IU every 6 h as a suspension
  Other Names: Mycostatin; Stamicin; Stamycin; Fungicidin; Nilstat
  Groups: Denture-related stomatitis group

SUMMARY:
The aim of this study is to evaluate the influence of presence of oral fungal infection, which leads to denture-related stomatitis, on blood pressure, endothelial function and immune cell phenotype in patients wearing dentures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dental prostheses used for at least 6 months,
* Substantial portion of the oral mucosa covered by dental prosthesis.

Exclusion Criteria:

* acute inflammatory disorders other than denture-related stomatitis, neoplastic disease relapses or chemotherapy courses less than 5 years before the enrolment,
* antibiotics in less than 4 weeks before the enrolment,
* anti-inflammatory drugs (steroids and non-steroidal, excluding aspirin in doses less than 80 mg) in less than 2 months before the enrolment,
* history of myocardial infarction, acute coronary incident or vascular inflammation in 5 weeks or less before the enrolment,
* chronic haematological disorders and immunodeficiencies less than 5 weeks before the enrolment,
* major medication changes less than 5 weeks before the enrolment or during study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dental clinic patients wearing dentures
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in blood pressure | Within 48h Prior to denture-related stomatitis treatment; 48h after recovery from denture-related stomatitis; 2 months after recovery from denture-related stomatitis
  Ambulatory Blood Pressure Monitoring System

SECONDARY OUTCOMES:
Change from baseline in endothelial function | Within 48h Prior to denture-related stomatitis treatment; 48h after recovery from denture-related stomatitis; 2 months after recovery from denture-related stomatitis
  Flow Mediated Dilatation
Changes in immune cell subset populations from baseline | Within 48h Prior to denture-related stomatitis treatment; 48h after recovery from denture-related stomatitis; 2 months after recovery from denture-related stomatitis
  Determination of cell subsets, activation markers and intracellular cytokine production

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Guzik, MD, PhD, Principal Investigator — Jagiellonian University; Marta Cześnikiewicz-Guzik, PhD, Principal Investigator — Jagiellonian University
Locations (2):
- Poland (2):
  - Zbigniew Żak Voivodeship Dental Clinic, Krakow
  - Jagiellonian University Dental Clinic, Krakow